CLINICAL TRIAL: NCT00690781
Title: Effect of Milk Proteins and Protein Feeding Pattern on Body Composition and Protein Metabolism in Energy Restricted Obese Subjects
Brief Title: Protein Nutrition During Weight Loss
Acronym: SURPROL-CF-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); ANRS, Emerging Infectious Diseases (Other Government); Université d'Auvergne (Other)
Responsible Party: Michel Beckert, Institut National de la Recherche Agronomique
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AU 724
Record Dates: First submitted 2008-05-30; First posted 2008-06-05 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Obesity
Keywords: casein; milk soluble proteins; protein feeding pattern; overweight; obesity; energy restriction; protein metabolism; lean body mass; body composition; nitrogen balance; protein synthesis; proteolysis; spread; pulse
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Casein Pulse (Experimental): casein is the main protein consumed, it is given during 6 weeks with a "pulse" protein feeding pattern : 8% for breakfast, 80% for lunch, 4% around 1600h, and 8% for dinner.
  Interventions: Dietary Supplement: Pulse casein feeding during energy restriction
- Casein Spread (Experimental): casein is the main protein consumed, it is given during 6 weeks with a "spread" protein feeding pattern : 25% for breakfast, 25% for lunch, 25% around 1600h, and 25% for dinner.
  Interventions: Dietary Supplement: Spread casein feeding during energy restriction
- MSP Pulse (Experimental): Milk soluble proteins (MSP) are the main protein consumed, it is given during 6 weeks with a "pulse" protein feeding pattern : 8% for breakfast, 80% for lunch, 4% around 1600h, and 8% for dinner.
  Interventions: Dietary Supplement: Pulse milk soluble protein feeding during energy restriction
- MSP Spread (Experimental): Milk soluble proteins (MSP) are the main protein consumed, it is given during 6 weeks with a "spread" protein feeding pattern : 25% for breakfast, 25% for lunch, 25% around 1600h, and 25% for dinner.
  Interventions: Dietary Supplement: Spread milk soluble protein feeding during energy restriction

INTERVENTIONS:
Dietary Supplement: Pulse casein feeding during energy restriction — Obese subjects are subjected to a 35% energy restriction during 6 weeks and during this period, 25% of energy is given as protein, these proteins being casein. In addition, a pulse protein feeding pattern is used (8% protein in the morning, 80% for lunch, 4% at 1600 h and 8% in the evening).
  Arms: Casein Pulse
Dietary Supplement: Spread casein feeding during energy restriction — Obese subjects are subjected to a 35% energy restriction during 6 weeks and during this period, 25% of energy is given as protein, these proteins being casein. In addition, a spread protein feeding pattern is used (25% of protein at each of the four meals of the day).
  Arms: Casein Spread
Dietary Supplement: Pulse milk soluble protein feeding during energy restriction — Obese subjects are subjected to a 35% energy restriction during 6 weeks and during this period, 25% of energy is given as protein, these proteins being milk soluble proteins. In addition, a pulse protein feeding pattern is used (8% protein in the morning, 80% for lunch, 4% at 1600 h and 8% in the evening).
  Arms: MSP Pulse
Dietary Supplement: Spread milk soluble protein feeding during energy restriction — Obese subjects are subjected to a 35% energy restriction during 6 weeks and during this period, 25% of energy is given as protein, these proteins being milk soluble proteins. In addition, a spread protein feeding pattern is used (25% of protein at each of the four meals of the day).
  Arms: MSP Spread

SUMMARY:
The purpose of this study is to minimize the loss of lean body mass that occurs during a weight-loss program in obese people by changing the nature of ingested protein and the pattern of protein feeding

DETAILED DESCRIPTION:
In most physiological situations, the adequate amount of protein necessary to promote health is more and more well known. However, for an adequate protein intake, it was shown that the kinetic of amino acid delivery to the organism has an influence on the efficiency of protein utilization. In particular, caseins, slowly digested milk proteins, promote a better protein balance than rapidly digested milk soluble proteins in young subjects (Boirie et al., 1997). In addition, changing protein feeding pattern (80% of daily protein consumed at noon vs 25%) significantly affect protein balance (Arnal et al., 2000). In young healthy individuals, the best protein efficiency is obtained by spreading protein absorption over time (casein, and/or 4 isoproteic meal per day). On the contrary, in older individuals, due to alteration in the sensitivity of protein metabolism to feeding, it is better to use rapidly digested proteins (Dangin et al., 2003), and / or to have a protein-rich meal once a day (Arnal et al., 1999).

Another physiological situation that was not studied in this regard is obesity. Obesity incidence is rapidly increasing around the world. When body mass index (weight / height2) becomes too high (>30), it is often suggested to restrict energy intake. However, severe energy restriction leads to fat mass loss, but also to lean body mass loss, which should be prevented. Our aim is to test whether for an adequate amount of total protein, it is possible to preserve lean body mass by using either casein, or milk soluble proteins, or by changing protein feeding pattern.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30
* sedentary
* normal TSH

Exclusion Criteria:

* any serious health problem

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Lean body mass | 6 weeks

SECONDARY OUTCOMES:
Nitrogen balance | 6 weeks
whole body leucine turnover | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, MD, Ph D, Professor, Principal Investigator — Université d'Auvergne, CHU de Clermont-Ferrand, Institut National de la Recherche Agronomique
Locations (1):
- Unité d'Exploration Nutritionnelle (Nutritional Exploration Unit), Clermont-Ferrand, France, France

REFERENCES:
- [Background] Arnal MA, Mosoni L, Boirie Y, Houlier ML, Morin L, Verdier E, Ritz P, Antoine JM, Prugnaud J, Beaufrere B, Mirand PP. Protein pulse feeding improves protein retention in elderly women. Am J Clin Nutr. 1999 Jun;69(6):1202-8. doi: 10.1093/ajcn/69.6.1202. PMID 10357740
- [Background] Arnal MA, Mosoni L, Boirie Y, Houlier ML, Morin L, Verdier E, Ritz P, Antoine JM, Prugnaud J, Beaufrere B, Mirand PP. Protein feeding pattern does not affect protein retention in young women. J Nutr. 2000 Jul;130(7):1700-4. doi: 10.1093/jn/130.7.1700. PMID 10867039
- [Background] Boirie Y, Dangin M, Gachon P, Vasson MP, Maubois JL, Beaufrere B. Slow and fast dietary proteins differently modulate postprandial protein accretion. Proc Natl Acad Sci U S A. 1997 Dec 23;94(26):14930-5. doi: 10.1073/pnas.94.26.14930. PMID 9405716
- [Background] Dangin M, Guillet C, Garcia-Rodenas C, Gachon P, Bouteloup-Demange C, Reiffers-Magnani K, Fauquant J, Ballevre O, Beaufrere B. The rate of protein digestion affects protein gain differently during aging in humans. J Physiol. 2003 Jun 1;549(Pt 2):635-44. doi: 10.1113/jphysiol.2002.036897. Epub 2003 Mar 28. PMID 12665610
- [Background] Dardevet D, Sornet C, Bayle G, Prugnaud J, Pouyet C, Grizard J. Postprandial stimulation of muscle protein synthesis in old rats can be restored by a leucine-supplemented meal. J Nutr. 2002 Jan;132(1):95-100. doi: 10.1093/jn/132.1.95. PMID 11773514
- [Background] Lacroix M, Bos C, Leonil J, Airinei G, Luengo C, Dare S, Benamouzig R, Fouillet H, Fauquant J, Tome D, Gaudichon C. Compared with casein or total milk protein, digestion of milk soluble proteins is too rapid to sustain the anabolic postprandial amino acid requirement. Am J Clin Nutr. 2006 Nov;84(5):1070-9. doi: 10.1093/ajcn/84.5.1070. PMID 17093159